CLINICAL TRIAL: NCT04029077
Title: Introduction in the NEtherlands of the Vapor Treatment for Patients With Severe Emphysema: a New Lungvolume Reduction Treatment
Brief Title: Introduction of the Vapor Treatment in The Netherlands
Acronym: NEVEL
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19 and other treatments available
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Pulmonary physician, University Medical Center Groningen
Other Study IDs: NEVEL-study
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Emphysema or COPD
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vapor group: Bronchoscopic lung volume reduction treatment using Vapor
  Interventions: Other: NA: intervention is not part of the study

INTERVENTIONS:
Other: NA: intervention is not part of the study — NA: it is not an interventional study

SUMMARY:
Rationale: The bronchoscopic lung volume reduction treatment using vapor was found to be effective and the treatment has an acceptable safety profile. The results of this trial has led to the inclusion of this treatment in the COPD GOLD guidelines in 2019. In the Netherlands the treatment has not been performed so far but the treatment device has been made available to the UMCG hospital to perform emphysema treatments. Some of the patients refered to the UMCG could benefit from the Vapor treatment and therefore with this treatment we will be able to treat patients who have no other treatment options left.

Objective: The overall aim of this study is to gain experience with the Thermal Vapor treatment by investigating the safety and efficacy of the treatment.

Primary Objective:

The primary objective is to investigate the change in Lung function (measured by Forced Expiratory Volume in 1 second (FEV1)) between baseline and 6 months after the Thermal Vapor treatment.

Study designThis study will be a prospective observational, single center study. All patients that undergo the bronchoscopic lung volume reduction treatment using thermal Vapor will be asked if their data can be captured in the database.

Study population: Patients with severe COPD who undergo the Thermal Vapor treatment.

DETAILED DESCRIPTION:
Rationale: The STEP-UP trial investigated the bronchoscopic lung volume reduction treatment using vapor and showed that the treatment group significantly improved after 6 months compared to the control group in Lung function and quality of life. The authors also concluded that the treatment has an acceptable safety profile. The results of this trial has led to the inclusion of this treatment in the COPD GOLD guidelines in 2019. In the Netherlands the treatment has not been performed so far but the treatment device has been made available to the UMCG hospital to perform emphysema treatments. Yearly, approximately 600 severe emphysema patients are refered to the UMCG for a bronchoscopic treatment but only approximately 10% is suitable for a treatment with endobronchial valves or coils. Some of the other patients could benefit from the Vapor treatment and therefore with this treatment we will be able to treat patients who have no other treatment options left.

Objective: The overall aim of this study is to gain experience with the Thermal Vapor treatment by investigating the safety and efficacy of the treatment.

Primary Objective:

The primary objective is to investigate the change in Lung function (measured by Forced Expiratory Volume in 1 second (FEV1)) between baseline and 6 months after the Thermal Vapor treatment.

Secondary Objectives:

Safety

• A secondary objective is to investigate the safety of the Thermal Vapor treatment by recoding all the adverse events that occur between baseline and 1 year follow up after treatment.

Efficacy • A secondary objective is to investigate the change in Lung function, lung hyperinflation, quality of life, dyspnea, CT parameters and exercise capacity between baseline and 6 and 12 months follow up after treatment.

Longterm

• A secondary objective is to investigate the long term effect of the treatment in terms of change in Lung function, lung hyperinflation, quality of life and exercise capacity between baseline and up to 5 years follow up after treatment.

Study designThis study will be a prospective observational, single center study that will investigate the safety and efficacy of the InterVapor (Bronchoscopic Thermal Vapor Ablation System) that will be introduced in the Netherlands for the first time. All patients that undergo the bronchoscopic lung volume reduction treatment using thermal Vapor will be asked if their data can be captured in the database.

Study population: Patients with severe COPD who undergo the Thermal Vapor treatment.

Main study parameters: The primary objective is to investigate the change in Lung function which will be measured by Forced Expiratory Volume in 1 second (FEV1) between baseline and 6 months after the Thermal Vapor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD
2. FEV1%pred <45% and FVC<70%pred,
3. Severe lung hyperinflation: RV>175%pred and RV/TLC>55%
4. Patients will have heterogeneous emphysema, as evidenced by high-resolution CT demonstrating a heterogeneity Index >1.2 in at least one segment to be treated.
5. Nonsmoking for at least 6 months prior to entering the study
6. Completed a pulmonary rehabilitation program within 6 months prior to treatment and/or regularly performing maintenance respiratory rehabilitation if initial supervised therapy occurred more than 6 months prior to baseline testing.
7. Read, understood and signed the Informed Consent form.

Exclusion Criteria:

1. FEV1 < 15% predicted
2. Inability to walk >140 meters in 6 minutes (6MWD) following optimized medical management
3. Subject has a history of recurrent clinically significant respiratory infections, defined as 3 or more hospitalizations for respiratory infection during the year prior to enrolment.
4. Highly diseased lower lobes (tissue to air ratio of <11%)
5. Presence of single large bulla (defined as > 1/3 volume of lobe) or a paraseptal distribution of emphysema in the treated lobe
6. Subject has severe pulmonary hypertension defined by right ventricular systolic pressure >45 mm Hg via echocardiogram.
7. Subject has severe gas exchange abnormalities as defined by: PaCO2 >8.0 kPa and/or PaO2 < 6.0 kPa (on room air).
8. Subject has an inability to tolerate bronchoscopy under conscious sedation or general anaesthesia.
9. Subject is taking >5 mg prednisone (or equivalent dose of a similar steroid) daily.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe COPD who undergo the Thermal Vapor treatment.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Lung function | Between baseline and 6 months follow up
  Change in Forced Expiratory Volume in 1 second (FEV1)

SECONDARY OUTCOMES:
Safety by number of adverse events | Between baseline and 1 year follow up
  Number of all adverse events
Lung function | Between baseline and 1 year follow up
  Change in Forced Expiratory Volume in 1 second
Hyperinflation | Between baseline and 6 months follow up
  Change in Residual Volume
Hyperinflation | Between baseline and 1 year follow up
  Change in Residual Volume
Quality of life measured by a questionnaire | Between baseline and 6 months follow up
  Change in St. George's Respiratory Questionnaire (SGRQ) total score (range 0-100, highest indicated worsed quality of life)
Quality of life measured by a questionnaire | Between baseline and 1 year follow up
  Change in St. George's Respiratory Questionnaire (SGRQ) total score (range 0-100, highest indicated worsed quality of life)
Exercise capacity | Between baseline and 6 months follow up
  Change in 6-minute walk distance (6MWD)
Exercise capacity | Between baseline and 12 months follow up
  Change in 6-minute walk distance (6MWD)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — Univeristy Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided
Only on request